CLINICAL TRIAL: NCT00961675
Title: A Phase III Clinical Study Evaluating the Efficacy Of FST-201 Otic Suspension (Foresight Biotherapeutics, Inc.) Vs. Ciprodex Otic Suspension (Alcon Laboratories, Inc.) in Subjects With Acute Otitis Externa
Brief Title: FST-201 in the Treatment of Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FST201-AOE-AS
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Acute Otitis Externa
Keywords: otitis; acute; externa; ear
MeSH Terms: conditions — Otitis | interventions — Dexamethasone; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FST201 (Active Comparator)
  Interventions: Drug: FST201 (dexamethasone 0.1% with povidone-iodine 1%)
- Ciprodex (Active Comparator)
  Interventions: Drug: Ciprodex (Ciprofloxacin 0.3%; dexamethasone 0.1% )

INTERVENTIONS:
Drug: FST201 (dexamethasone 0.1% with povidone-iodine 1%) — 4 gtt BID (twice a day)
  Arms: FST201
Drug: Ciprodex (Ciprofloxacin 0.3%; dexamethasone 0.1% ) — 4 gtt BID (twice a day)
  Other Names: CIPRODEX® (ciprofloxacin 0.3% and dexamethasone 0.1%) Sterile Otic Suspension
  Arms: Ciprodex

SUMMARY:
The objective of this study is to evaluate the efficacy of FST-201 compared to Ciprodex in the treatment of acute otitis externa. This study will be conducted at one site, the Lyndon B. Johnson (LBJ) Tropical Medical Center, Department of Otolaryngology, in Pago Pago, American Samoa.

DETAILED DESCRIPTION:
The proposed clinical trial will evaluate the efficacy of FST-201 (dexamethasone 0.1% with povidone-iodine 1% ) Otic Suspension vs. the FDA-approved drug Ciprodex (ciprofloxacin 0.3%, dexamethasone 0.1%) Otic Suspension (Alcon Laboratories, Inc.) in the treatment of acute otitis externa. Acute otitis externa is a common inflammatory condition of the external auditory canal often associated with infection, allergy and dermatitis. The active ingredient in our novel dexamethasone suspension is identical in concentration and route of administration to the steroid component of the approved drug Ciprodex, which is currently the most widely-prescribed dexamethasone-containing agent in the treatment of acute otitis externa. We will enroll 60 patients (30 each in two separate treatment groups) in this trial. All patients electing to participate in this study will receive either FST-201 or Ciprodex. FST-201 and Ciprodex will be masked and provided free of charge to all study participants. Patients will be followed for at least 15 days or until their ear inflammation is either resolved or determined to need additional interventions. The study will be conducted with attention to all relevant Good Clinical Practice (GCP), International Conference on Harmonization (ICH), FDA, Health Insurance Portability and Accountability Act (HIPPA) and Declaration of Helsinki guidelines.

ELIGIBILITY:
Inclusion Criteria:

Study participants must:

* Have a clinical diagnosis of AOE in one or both ears, defined as a clinical score of at least 1 for edema (0-3 scale), 2 for overall inflammation (0-3 scale) and 1 for tenderness (absent=0, present=1)
* Be at least 18 years of age at Visit 1 (Day 1, Screening/Baseline) of either sex and any race

Exclusion Criteria:

Study participants must NOT:

* Have known sensitivity to any component of the study medications
* Have a current infection requiring systemic antimicrobial treatment
* Have used topical or systemic pain meds on the same day as Screening/Baseline Visit 1 and for the duration of the study.
* Take any systemic (within 30 days) or otic corticosteroids (within 1 days) prior to Screening/Baseline Visit 1
* Current use of topical or systemic non-steroidal or other anti-inflammatory drugs
* Use any topical otic treatment with alcohol, vinegar, hydrogen peroxide or other astringent medication during the course of the study or on the same day as Screening/Baseline Visit 1
* Have taken any antibiotics within 3 days prior to Visit 1
* Have signs and symptoms of AOE for > 4 weeks at Screening/Baseline Visit 1
* Have a clinical diagnosis of malignant otitis externa;
* Have overt fungal AOE
* Have a viral infection of the pinna or tympanic membrane (i.e herpes zoster)
* Have congenital abnormalities of the external auditory canal in the enrolled ear(s)
* Have obstructive bony exostoses in the enrolled ear(s);
* Have mastoid or other suppurative, non-infectious ear disorders (e.g, cholesteatoma)
* Have malignant tumors of the external auditory canal
* Have a history of otologic surgery. Surgery performed more than 1 year prior to Screening/Baseline Visit 1and limited to the tympanic membrane is allowed
* Have seborrheic dermatitis of the external auditory canal
* Have a current or prior history of immunosuppressive disorders
* Be pregnant, nursing or planning a pregnancy

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Overall clinical cure as defined by absence of the signs and symptoms of Acute Otitis Externa (AOE) including ear inflammation, edema, tenderness and otic discharge. | 18 days

SECONDARY OUTCOMES:
Microbiological resolution defined as elimination of pre-treatment pathogenic organism. | 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- LBJ Tropical Medical Center, Department of Otolaryngology, Pago Pago, American Samoa